CLINICAL TRIAL: NCT06727682
Title: Feasibility and Relevance of Stress Management Education Delivered Via Virtual Classroom for Carers Working in Specialised Care Units in Nursing Homes: a Pilot Study of a Randomized Controlled Trial
Brief Title: Feasibility of Stress Management Education Delivered Via Virtual Classroom in Nursing Homes: a Pilot Study of a RCT
Acronym: AGIT-RESTS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS CIPS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AGIT-RESTS-1
Record Dates: First submitted 2024-11-29; First posted 2024-12-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Occupational Stress
Keywords: stress management; virtual classroom; risk of burnout; behavioural and psychological symptoms of dementia
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Cluster-randomised pilot study with four specialised care units of nursing homes and two clusters. Two specialised care units will be randomized in the experimental cluster, and the other ones will be randomized in the control cluster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote stress management programme (Experimental): Ten-hour, three-course stress management programme with a psychologist via video conferencing over 2 months
  Interventions: Behavioral: Stress management
- Waiting list (No Intervention): No intervention during the study duration. However, after the end of the study, after the last evaluations, participants in this control cluster will be offered the opportunity to follow the stress management programme.

INTERVENTIONS:
Behavioral: Stress management — Ten-hour, three-course stress management programme with a psychologist via video conferencing over a 2 month period. The classes will be delivered in small groups of maximum seven care workers. Carers can be brought together in the same room, but the speaker will necessarily be at a distance, via videoconferencing. The formation will adress the following issues: i) Understanding the mechanisms of stress, ii) Identifying sources of stress and triggers, iii) Anticipate stressful situations and use their resources to prevent them, and iv) Use the most appropriate stress-reduction techniques, depending on their sensitivity.
  Arms: Remote stress management programme

SUMMARY:
The aim of this cluster-randomised pilot study is to assess the feasibility of a remote stress management programme to reduce occupational stress in healthcare workers in specialised care units of nursing homes. Secondary aims are to assess the effectiveness of the programme in reducing stress in care workers and reducing behavioural and psychological symptoms of dementia in residents.

Participants randomised to the experimental cluster will follow the stress management programme delivered in a virtual classroom. Participants randomised to the control cluster will be placed on a waiting list.

The primary outcome measure will be the participation rate in the study. Other secondary outcomes will include measures of heart rate variability (as a marker of physiological stress) and scores on specific questionnaires for stress, anxiety and risk of burnout in nursing staff in the specialised care units, and behavioural and psychological symptoms of dementia and quality of life in residents in the specialised care units.

Both clusters will complete the same assessments. Participants in the experimental cluster will follow a three-course programme with a psychologist via videoconferencing over a period of 2 months. After the study's final evaluation visit, which will take place one month after the programme, participants in the control cluster will be offered the opportunity to follow the same programme.

ELIGIBILITY:
Inclusion Criteria:

* Having a caring relationship with residents (e.g. nurses, nursing assistants)
* Working in the specialised care unit of the nursing home
* Working in the nursing home for at least 3 months on the date of inclusion and whose employment contract does not end within 3 months of the date of inclusion.
* Obtaining express written informed consent, after a period of reflection

Exclusion Criteria:

* Person in a period of relative exclusion in relation to another protocol
* Person who is not affiliated to or does not benefit from a social security scheme.
* Pregnant or lactating woman
* Participant unable to give consent
* Person deprived of liberty by judicial or administrative decision
* Person unable to understand, speak, read and write French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Participation rate | From enrollment to the end of the study at 3 months
  Participation rate defined as the ratio of the number of participants who completed all study visits to the number of care professionals who agreed to participate.

SECONDARY OUTCOMES:
Acceptance rate | At enrollment
  Ratio between the total number of eligible healthcare workers and the number of healthcare worker who accept to be enrolled in the study.
Retention rate | From enrollment to the end of the study at 3 months
  Ratio between the number of care professionals still present at the last visit of the study and the number of care professionals included in the study
Adherence | From the beginning to the end of the study, at 3 months
  Average number of visits attended by each participant.
Quality of the intervention | At the end of the intervention, at 3 months
  Feedback on the relevance of the training and its contribution through semi-directive interviews and focus groups in participants and in managers and directors of the nursing homes.
Cost of the programme | From enrollment to the end of the study at 3 months
  Total cost of the stress management program including the costs incurred to enable the employee to follow the training and/or the costs incurred to replace the absence of the employee in the service
Heart rate variability | Baseline and 3 months
  Recording of resting heart rate variability assessed by RMSSD, SDNN, LF and HF markers.
Occupational stress | Baseline, 2 months and 3 months
  Score on the Work Place Stress Scale
Overall stress | Baseline, 2 months and 3 months
  Score on the Perceived Stress Scale-10
Job satisfaction | Baseline, 2 months and 3 months
  Score on the Overall Job Satisfaction Scale
Risk of burn-out | Baseline, 2 months and 3 months
  Score on the Malasch Burnout Inventory
Quality of life | Baseline, 2 months and 3 months
  Score on the World Health Organization Quality of Life questionnaire
Self-rated health | Baseline, 2 months and 3 months
  Score on the self-rated health scale
Anxiety | Baseline, 2 months and 3 months
  Score on the Generalized Anxiety Disorder 7-Item
Perceptions of the quality of patient care | Baseline, 2 months and 3 months
  Score on the Victorian Patient Satisfaction Questionnaire
Substance use | Baseline, 2 months and 3 months
  Usual substance use (tobacco, alcohol, drugs...), assessed by a questionnaire that records the type of substance and frequency of use.
Knowledge and mastery of stress management tools | Baseline, 2 months and 3 months
  Score on a multiple-choice questionnaire specially designed for the study

OTHER OUTCOMES:
Residents' level of agitation in the specialised care units | Baseline and 3 months
  Perceived residents' level of agitation by the healtcare workers assessed by the score on the Cohen-Mansfield Agitation Inventory
Health-related quality of life of residents in the specialised care units | Baseline and 3 months
  Residents' health-related quality of life as perceived by healthcare workers, as assessed by scores on the 'Quality of Life in Late Stage Dementia' questionnaire.
Behavioural and psychological symptoms of dementia in the residents of the specialised care units | Baseline and 3 months
  Residents' behavioural and psychological symptoms of dementia as perceived by healthcare workers, as assessed by the "Neuropsychiatric inventory" questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Kabirian, MD, Principal Investigator — France Chief Medical Officer, Clariane
Locations (4):
- France (4):
  - Korian La Colombe, Gigean, France
  - Korian Le Clos de l'orchidée, Narbonne, Occitanie
  - Korian Parc de l'abbaye, Saint-Cyr-l'École, Île-de-France Region
  - Korian Parc des dames, Saint-Germain-en-Laye, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided